CLINICAL TRIAL: NCT00658216
Title: Usefulness of Measuring Plasma Brain Natriuretic Peptide for Diagnosis and Prognosis in Very Elderly Patients.
Brief Title: Brain Natriuretic Peptide (BNP) Usefulness In Elderly Dyspneic Patients (BED)
Acronym: BED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: SCR 06 007
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: Diagnosis and prognosis; Very elderly population; Heart failure; Brain natriuretic peptide; Observational prospective study; Older; Dyspneic patients aged 80
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for brain natriuretic peptide measurement
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Longitudinal: Prospective study : cohort of consecutive patients recruited over 2 years

SUMMARY:
The purpose of this study is to test the usefulness of measuring plasma brain natriuretic peptide (BNP) for diagnosis and prognosis in very elderly dyspneic patients.

DETAILED DESCRIPTION:
Measurement of BNP concentration is approved for use in the diagnosis of heart failure (HF) in elderly patients below 80 years of age. The value of plasma BNP assays as diagnostic tools has not been determined in very elderly populations because the plasma BNP increases with age. This large, multicenter, prospective, observational, study in 300 participants is aimed to prospectively test the usefulness of measuring plasma BNP for diagnosis of HF in dyspneic patients aged 80 and older.

ELIGIBILITY:
Inclusion Criteria:

* acute dyspnea
* crackles on lung auscultation,
* hypoxemia,
* right-sided signs.

Exclusion Criteria:

* no exclusion criteria

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Defined population
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Plasma BNP levels at T0 to test the optimal values of measuring plasma BNP for diagnosis of HF in patients older than 80 years. | 6 months

SECONDARY OUTCOMES:
Plasma BNP levels at 3 times (T0, T48, Tend) to test the usefulness of measuring plasma BNP : 1.at T0 : in diagnosing HF using a 2-threshold up-and down-approach | 6 months
2.at T48 : in diagnosing and prognosing HF using a 2nd assay after 48 hours of treatment | 6 months
3.at Tend : in prognosing HF using a 3rd assay after the acute phase (composite criteria) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Broca Hospital, Paris, France

REFERENCES:
- [Background] Komajda M, Hanon O, Aupetit JF, Benetos A, Berrut G, Emeriau JP, Friocourt P, Galinier M, De Groote P, Jondeau G, Jourdain P, Forette F. Management of heart failure in the elderly: recommendations from the French Society of Cardiology (SFC) and the French Society of Gerontology and Geriatrics (SFGG). J Nutr Health Aging. 2006 Sep-Oct;10(5):434-44. PMID 17066218
- See also: The French Society of Cardiology (SFC) — http://www.sfcardio.fr/
- See also: the French Society of Gerontology and Geriatrics (SFGG). — http://www.sfgg.fr/